CLINICAL TRIAL: NCT02011698
Title: Absorbable Sutures , Non Absorbable Sutures or Biologic Fibrin Glue for Protesic Mesh Fixing in Lichtenstein Technique for Primitive Groin Hernia Repair: a Randomized Prospective Multicentric Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale di Circolo - Fondazione Macchi (Other)
Responsible Party: Principal Investigator, Lorenzo Latham, MD, MD, Ospedale di Circolo - Fondazione Macchi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Hernia-01
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Hernia, Inguinal
Keywords: Groin hernia; lichtenstein herniorrhaphy
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- absorbable sutures (Experimental): mesh fixation with absorbable sutures in lichtenstein anterior inguinal herniorrhaphy
  Interventions: Procedure: Lichtenstein technique groin hernia repair with mesh. Use of absorbale sutures for mesh fixation
- non absorbable sutures (Active Comparator): mesh fixation with non absorbable sutures in lichtenstein anterior inguinal herniorrhaphy. This is the method to be considered the standard of care thus far.
  Interventions: Procedure: Lichtenstein technique groin hernia repair with mesh. Use of non absorbable sutures for mesh fixation
- fibrin biological glue (Experimental): mesh fixation with fibrin biological glue in lichtenstein anterior inguinal herniorrhaphy
  Interventions: Procedure: Lichtenstein technique groin hernia repair with mesh. Use of fibrin biological glue for mesh fixation

INTERVENTIONS:
Procedure: Lichtenstein technique groin hernia repair with mesh. Use of absorbale sutures for mesh fixation
  Arms: absorbable sutures
Procedure: Lichtenstein technique groin hernia repair with mesh. Use of non absorbable sutures for mesh fixation
  Arms: non absorbable sutures
Procedure: Lichtenstein technique groin hernia repair with mesh. Use of fibrin biological glue for mesh fixation
  Arms: fibrin biological glue

SUMMARY:
this study has the aim to analize the correlation between three different methods of mesh fixation ( using absorbable or non absorbable sutures or fibrin biological glue) and recurrance and chronic pain ,in the Lichtenstein anterior inguinal erniorrhaphy

DETAILED DESCRIPTION:
In the last decades the rate of recurrence in the anterior inguinal erniorraphy has been drastically lowered with the introduction of the mesh , on the other hand the rate of chronic pain is reported to be high in many papers.

The chronic pain influences the quality of life and what's more causes an increase in the social costs.

the classical Lichtenstein inguinal anterior erniorrhaphy , wich is the technique suggested by the international guidelines, expected to fix the mesh with non absorbable sutures .

The investigators would analyze the possible correlation between the method of mesh fixation and chronic pain keeping a lower rate of recurrence.

That said the primary endpoint in this study is the rate of recurrence and the secondary endpoint is the rate of chronic pain after lichtenstein anterior inguinal erniorrhaphy in the three different methods of fixation of the mesh

ELIGIBILITY:
Inclusion Criteria:

* primitive inguinal hernia
* age > 18 years old
* compliancy to the study

Exclusion Criteria:

* reccurent inguinal hernia
* age < 18 years old
* refusal of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
rate of recurrence | 1 year

SECONDARY OUTCOMES:
rate of chronic pain | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Latham, MD, Principal Investigator — Department of Surgery. Azienda Ospedaliera Ospedale di Circolo e Fondazione Macchi; Eugenio Cocozza, MD, Study Director — Department of Surgery. Azienda Ospedaliera Ospedale di Circolo e Fondazione Macchi; Lorenzo Livraghi, MD, Principal Investigator — Department of Surgery. Azienda Ospedaliera Ospedale di Circolo e Fondazione Macchi; Mattia Berselli, MD, Principal Investigator — Department of Surgery. Azienda Ospedaliera Ospedale di Circolo e Fondazione Macchi; Bianca Gambitta, Student, Study Chair — Department of Surgery. Azienda Ospedaliera Ospedale di Circolo e Fondazione Macchi; Luca Farassino, MD, Study Chair — Department of Surgery. Azienda Ospedaliera Ospedale di Circolo e Fondazione Macchi; Ildo Scandroglio, MD, Study Chair — Department of surgery Azienda Ospedaliera di Busto Arsizio Ospedale di Tradate; Francesco Roscio, MD, Study Chair — Department of surgery Azienda Ospedaliera di Busto Arsizio ospedale di Tradate; Dario Maggioni, MD, Study Chair — Azienda Ospedaliera, Ospedale Civile di Legnano; Angelo Miranda, MD, Study Chair — Azienda Ospedaliera, Ospedale Civile di Legnano
Locations (1):
- Azienda Ospedaliera Ospedale di Circolo e Fondazione Macchi, Varese, Va, Italy

REFERENCES:
- [Background] Dick AC, Deans GT, Irwin ST. A prospective study of adult inguinal hernia repairs using absorbable sutures. J R Coll Surg Edinb. 1996 Oct;41(5):319-20. PMID 8908956
- [Background] Paajanen H. Do absorbable mesh sutures cause less chronic pain than nonabsorbable sutures after Lichtenstein inguinal herniorraphy? Hernia. 2002 Mar;6(1):26-8. doi: 10.1007/s10029-002-0048-2. PMID 12090577
- [Background] Holzheimer RG. Inguinal Hernia: classification, diagnosis and treatment--classic, traumatic and Sportsman's hernia. Eur J Med Res. 2005 Mar 29;10(3):121-34. PMID 15851379
- [Background] de Goede B, Klitsie PJ, van Kempen BJ, Timmermans L, Jeekel J, Kazemier G, Lange JF. Meta-analysis of glue versus sutured mesh fixation for Lichtenstein inguinal hernia repair. Br J Surg. 2013 May;100(6):735-42. doi: 10.1002/bjs.9072. Epub 2013 Feb 22. PMID 23436683
- See also: Related Info — http://www.ssat.com/cgi-bin/hernia6.cgi